CLINICAL TRIAL: NCT03593213
Title: A Double-Blind, Placebo-Controlled, Randomized Withdrawal, Multicenter Clinical Trial Evaluating the Efficacy, Safety, and Tolerability of Cariprazine in a Dose-Reduction Paradigm in the Prevention of Relapse in Patients With Schizophrenia
Brief Title: Clinical Trial Evaluating the Efficacy, Safety, and Tolerability of Cariprazine in a Dose-Reduction Paradigm in the Prevention of Relapse in Participants With Schizophrenia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: FDA Released Allergan from this post marketing requirement
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RGH-MD-24; 2017-000818-34 (EudraCT Number); NCT04519099 (obsolete NCT alias)
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Results first posted 2022-03-08 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — cariprazine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cariprazine 4.5 mg/day (Open-label Treatment Period) (Experimental): Cariprazine 1.5 mg capsules orally once daily at Week 1, titrated to 3.0 mg capsules orally once daily at Week 2 and then titrated to 4.5 mg orally once daily from Week 3 through Week 18 in the Open-label Treatment Period.
  Interventions: Drug: Cariprazine
- Placebo (Double-blind Treatment Period) (Placebo Comparator): Cariprazine placebo-matching capsules orally once daily from Week 19 through Week 44 in Double-blind Treatment Period.
  Interventions: Drug: Placebo
- Cariprazine 3.0 mg/day (Double-blind Treatment Period) (Experimental): Cariprazine 3.0 mg capsules orally once daily from Week 19 through Week 44 in Double-blind Treatment Period.
  Interventions: Drug: Cariprazine
- Cariprazine 4.5 mg/day (Double-blind Treatment Period) (Experimental): Cariprazine 4.5 mg capsules orally once daily from Week 19 through Week 44 in Double-blind Treatment Period.
  Interventions: Drug: Cariprazine

INTERVENTIONS:
Drug: Cariprazine — Cariprazine capsules, oral administration, once daily.
  Arms: Cariprazine 3.0 mg/day (Double-blind Treatment Period); Cariprazine 4.5 mg/day (Double-blind Treatment Period); Cariprazine 4.5 mg/day (Open-label Treatment Period)
Drug: Placebo — Matching placebo capsules, oral administration, once daily.
  Arms: Placebo (Double-blind Treatment Period)

SUMMARY:
1. To evaluate the efficacy and safety of cariprazine at a target dose of 4.5 milligram per day (mg/d) compared with placebo in prevention of relapse in patients with schizophrenia
2. To evaluate the efficacy and safety of cariprazine at a target dose of 3.0 mg/d compared with placebo in prevention of relapse in patients with schizophrenia who were initially stabilized on a target dose of 4.5 mg/d

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia for a minimum of 1 year before Visit 1 (Screening).
* Ability to follow study instructions, complete study assessment tools with minimal assistance and no alteration to the assessment tools, and likely to complete all required visits.
* Participant meets Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for schizophrenia as determined by Structured Clinical Interview for DSM-5 (SCID-5).
* Positive and Negative Syndrome Scale (PANSS) total score >= 70 and <= 120 at Visit 1 and Visit 2 (Day 1).
* Rating of at least 4 (moderate) on at least 2 of the following 4 PANSS positive symptoms; P1: delusions; P2: conceptual disorganization; P3: hallucinatory behaviour; P6: suspiciousness/persecution at Visit 1 and Visit 2.

Exclusion Criteria:

* Currently meeting DSM-5 criteria for any of the following:
* Schizoaffective disorder, schizophreniform disorder, and other psychotic disorders
* Bipolar I and II disorder
* Autism spectrum disorder, intellectual development disorder, delirium, major/minor neurocognitive disorder
* History of meeting DSM-5 criteria for substance-related disorders (excluding caffeine-related and tobacco-related disorders) within the prior 3 months before Visit 1.
* Prior participation in any clinical trials involving experimental or investigational drugs within 6 months before Visit 1 or planned during the study.
* Female Participants who are pregnant, planning to become pregnant during the course of the study, or are currently lactating.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 587 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-02-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (96):
- United States (42):
  - Pillar Clinical Research, Bentonville, Arkansas
  - Woodland International Research Group, Little Rock, Arkansas
  - Woodland Research Northwest, LLC, Rogers, Arkansas
  - Advanced Research Center, Inc., Anaheim, California
  - CITrials - Bellflower, Bellflower, California
  - Synexus Clinical Research US, Inc., Cerritos, California
  - ATP Clinical Research, Inc., Costa Mesa, California
  - California Pharmaceutical Research Institute, Inc., Costa Mesa, California
  - ProScience Research Group, Culver City, California
  - Collaborative Neuroscience Research Network, LLC., Garden Grove, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Omega Clinical Trials, La Habra, California
  - Synergy San Diego, Lemon Grove, California
  - Alliance Research, Long Beach, California
  - Excell Research, Inc, Oceanside, California
  - Orange County Neuropsychiatric Research Center, LLC, Orange, California
  - CNRI-Los Angeles, Pico Rivera, California
  - University of California San Diego, San Diego, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Collaborative Neuroscience Research, LLC, Torrance, California
  - Wilks & Safirstein MD PA D/B/A MD Clinical, Hallandale, Florida
  - Southern Winds Hospital, Hialeah, Florida
  - Research Centers of America, Hollywood, Florida
  - Synexus Clinical Research, Inc, Atlanta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta LLC, Decatur, Georgia
  - Atlanta Behavioral Research, LLC, Dunwoody, Georgia
  - AMITA Health Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - Louisiana Clinical Research, Shreveport, Louisiana
  - CBH Health LLC, Gaithersburg, Maryland
  - Altea Research, Las Vegas, Nevada
  - Alea Research Institute, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - New Hope Clinical Research, Charlotte, North Carolina
  - Clinical Inquest Center Ltd., Beavercreek, Ohio
  - OSY Psychiatry Department, Columbus, Ohio
  - Professional Psychiatric Services, Mason, Ohio
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Community Clinical Research, Inc., Austin, Texas
  - Pillar Clinical Research, Richardson, Texas
  - Pillar Healthcare, Richardson, Texas
- Bulgaria (10):
  - Mental Health Centre - Prof.Dr.Ivan Temkov-Burgas, Burgas
  - State Psychiatry Hospital, Kardzhali
  - MHAT Dr. Hristo Stambolski" EOOD; Department of Psychiatry, Kazanlak
  - State Psyciiatric Hospital - Lovech, Lovech
  - UMHAT Dr. Georgi Stranski, EAD, Pleven
  - Mental health Centre-Ruse EOOD, Rousse
  - MHAT-Targovishte, AD, Targovishte
  - DCC Mladost M - Varna, OOD, Varna
  - Mental Health Center - Veliko Tarnovo EOOD, Veliko Tarnovo, Veliko Tarnovo
  - Mental Health Center - Vratsa EOOD, Vratsa, Vratsa
- Malaysia (3):
  - University Kuala Lumpur, Ipoh
  - University Malaya Medical Center, Kuala Lumpur
  - Hospital Sentosa, Kuching
- Poland (5):
  - Szpital Uniwersytecki Nr.1 im. Dr. A. Jurasza, Klinika Psychiatrii, Bydgoszcz
  - Samodzielny Publiczny Zespół Opieki Zdrowotnej, Chełmno
  - Centrum Badan Klinicznych PI-House, Gdansk
  - Specjalistyczna Praktyka lekarska, Lublin
  - Indywidualna Specjalistyczna Praktyka, Poznan
- INSPIRA Clinical Research, San Juan, Puerto Rico
- Romania (5):
  - Spitalul de Psihiatrie si Neurologie Brasov, Brasov
  - Spitalul de Psihiatrie TITAN "Dr. Constantin Gorgoș", Bulevardul Nicolae Grigorescu, Nr. 41, Bucharest
  - Armys Clinical Emergency Central Hospital Prof Dr Carol Davila, Bucharest
  - CETTT SF Stelian Hospital, Bucharest
  - Spital Clinic Judetean Tg. Mures, Târgu Mureş
- Serbia (7):
  - Clinical Center of Serbia, Belgrade
  - Clinical Hospital Center Dr. Dragisa Misovic-Dedinje, Belgrade
  - Institute of Mental Health, Belgrade
  - Special Hospital for Psychiatric Diseases "Kovin", Kovin
  - Clinical Centre Kragujevac, Kragujevac
  - Specialized Hospital for Neuropsychiatric Diseases Sveti Vracevi, Novi Kneževac
  - Clinic for Psychiatry, Clinical Centre of Vojvodina, Novi Sad
- South Korea (5):
  - Inje University Busan Paik Hospital, Busan
  - Inje University Heaundae Paik Hospital, Busan
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Jeju National University Hospital, Jeju City
- Taiwan (3):
  - Taipei Tzu Chi Hospital, New Taipei City
  - National Cheng Kung University Hospital, Tainan
  - Department of Psychiatry, Taipei Veterans General Hospital, Taiwan, Taipei
- Suan prung Psychiatric Hospital, Nonthaburi, Thailand
- Ukraine (14):
  - Regional Psychonevrological Hospital #3, Ivano-Frankivsk
  - Kharkiv regional clinical psychiatric hospital #3, Kharkiv
  - Institute of Neurology, Psychiatry and Narcology of the NAMS of Ukraine, Kharkiv
  - SI Institute of Neurology, Psychiatry and Narcology of NAMSU, Kharkiv
  - Kyiv Railway Clinical Hospital #2 of Branch "Health Center" of the Public Joint Stock Company "Ukrainian Railway"v, Kyiv
  - Kyiv Regional Medical Incorporation "Psychiatry", Kyiv
  - Geikivka multidisciplinary hospital for psychiatric care, Kyiv
  - KNP of Lviv Regional Council "Lviv Regional Clinical Psychiatric Hospital", Lviv
  - Odessa Regional Medical Centre of Mental Health, Odesa
  - Odesa Regional Psychiatric Hospital No.2 of the ORC, Odesa
  - Kherson Regional Psychiatric Institution for Psychiatric Care, Petrivka
  - Cherkasy regional psychiatric hospital of the CRC, Smila
  - CI O.I. Yuschenko VRPsH Depts No.14 and No.15 M.I. Pyrogov VNMU, Vinnytsia
  - VNMU, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Period: Open-label Treatment Period (18 Weeks)
Arm/Group | Cariprazine 4.5 mg/Day (Open-label Treatment Period) | Placebo (Double-blind Treatment Period) | Cariprazine 3.0 mg/Day (Double-blind Treatment Period) | Cariprazine 4.5 mg/Day (Double-blind Treatment Period)
Started | 587 (Out of 162 participants who completed Open-label Treatment Period, 159 participants were randomized to Double-blind treatment Period.) | 0 | 0 | 0
Completed | 162 | 0 | 0 | 0
Not Completed | 425 | 0 | 0 | 0
Not completed — Adverse Event | 39 | 0 | 0 | 0
Not completed — Lack of Efficacy | 14 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 85 | 0 | 0 | 0
Not completed — Lost to Follow-up | 51 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Protocol Deviation | 5 | 0 | 0 | 0
Not completed — Non-compliance with Study Drug | 23 | 0 | 0 | 0
Not completed — Study Terminated by the Sponsor | 90 | 0 | 0 | 0
Not completed — Reason not Specified | 13 | 0 | 0 | 0
Not completed — Failure to Meet Randomization Criteria | 104 | 0 | 0 | 0
Period: Double-blind Treatment Period (26 Weeks)
Arm/Group | Cariprazine 4.5 mg/Day (Open-label Treatment Period) | Placebo (Double-blind Treatment Period) | Cariprazine 3.0 mg/Day (Double-blind Treatment Period) | Cariprazine 4.5 mg/Day (Double-blind Treatment Period)
Started | 0 | 54 | 49 | 56
Safety Population (Double-blind Safety Population included all participants who took at least 1 dose of cariprazine during and double-blind treatment period.) | 0 | 53 | 49 | 54
Completed | 0 | 14 | 16 | 21
Not Completed | 0 | 40 | 33 | 35
Not completed — Number of Participants with Relapse Event | 0 | 15 | 9 | 8
Not completed — Adverse Event | 0 | 2 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 4 | 2 | 3
Not completed — Lost to Follow-up | 0 | 5 | 4 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Protocol Deviation | 0 | 3 | 2 | 5
Not completed — Non-compliance with Study Drug | 0 | 1 | 2 | 0
Not completed — Study Terminated by Sponsor | 0 | 9 | 11 | 13
Not completed — Reason not Specified | 0 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Double-blind Safety Population included all participants who took at least 1 dose of cariprazine during and double-blind treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Double-blind Treatment Period) | Cariprazine 3.0 mg/Day (Double-blind Treatment Period) | Cariprazine 4.5 mg/Day (Double-blind Treatment Period) | Total
Number analyzed (Participants) | 53 | 49 | 54 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (10.94) | 40.6 (10.84) | 42.7 (11.08) | 41.7 (10.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 22 | 53
  Male | 39 | 32 | 32 | 103
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 34 | 38 | 39 | 111
  White | 17 | 11 | 11 | 39
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 10 | 12 | 10 | 32
  Non-Hispanic | 43 | 37 | 44 | 124

OUTCOME MEASURES:

1. Primary Outcome: Time to First Relapse During Double-blind Treatment Period
Description: Time to Relapse is the number of days from randomization to first relapse.
  Relapse is defined as any 1 of the following:
  * Increase in Positive and Negative Syndrome Scale(PANSS) by ≥30% for participants who had total score of ≥50 at randomization or ≥10-point increased score with total score <50 at randomization [PANSS=30 questions where 1=absence of symptoms to 7=extremely severe symptom;total score=30 to 210;higher score more severe symptoms]
  * Increase in Clinical Global Impression-Severity (CGI-S) score by 2 or more points [1=normal to 7=among most extremely ill]
  * Score of >4 on 1 or more of 7 PANSS items:P1-delusions,P2-conceptual disorganization,P3-hallucinatory behavior,P6-suspiciousness,P7-hostility,G8-uncooperativeness,G14-poor impulse control
  * Deliberate self-injury
  * Initiation of treatment with mood stabilizer,antidepressant,antipsychotics or benzodiazepine that exceeds specified allowance
  * Psychiatric hospitalization
  * Exacerbation of psychiatric illness
Time Frame: Randomization (Week 18) to End of Treatment (Week 44)
Population: The Double-blind Intent-to Treat (DB ITT) population included all participants in the DB safety population who had at least 1 post-randomization assessment of the PANSS or CGI-S scores during the DB treatment period of the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo (Double-blind Treatment Period) | Cariprazine 3.0 mg/Day (Double-blind Treatment Period) | Cariprazine 4.5 mg/Day (Double-blind Treatment Period)
Number analyzed (Participants) | 53 | 49 | 53
days | NA [183.0 to NA] — The median, and upper limit of 95% confidence interval (CI) was not estimable due to low number of participants with event. | NA [184.0 to NA] — The median, and upper limit of 95% CI was not estimable due to low number of participants with event. | NA [NA to NA] — The median, lower and upper limit of 95% CI was not estimable due to low number of participants with event.
Statistical Analysis 1: Comparison: Placebo (Double-blind Treatment Period) vs Cariprazine 3.0 mg/Day (Double-blind Treatment Period); Test type: Superiority; p = 0.1576, Log Rank — The significance level was 0.05 using the log rank test; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.25 to 1.29] — Hazard ratio (cariprazine 3.0 or 4.5 mg/day vs. placebo) was based on Cox proportional hazards regression model, with treatment group as an explanatory variable
Statistical Analysis 2: Comparison: Placebo (Double-blind Treatment Period) vs Cariprazine 4.5 mg/Day (Double-blind Treatment Period); Test type: Superiority; p = 0.2066, Log Rank — The significance level was 0.05 using the log rank test; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.26 to 1.45] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: First dose to last dose + 30 days in the Open-label Treatment Period (Up to 23 weeks); First dose to last dose + 30 days in the Double-blind Treatment Period (Up to 35 weeks)
Description: All-cause mortality included all participants. Open-label (OL) Safety Population (OLTP) included all participants in the screened population who took at least 1 dose of OL cariprazine during the OLTP of the study. DB safety population included all participants in the randomized population who took at least 1 dose of DB IP.
Groups:
- Cariprazine 4.5 mg/Day (Open-label Safety Follow-up): Safety Follow-up Period following treatment with Cariprazine 4.5 mg/day in the Open-label Treatment Period for participants who did not continue to the Double-blind Treatment Period.
- Placebo (Double-blind Safety Follow-up): Safety Follow-up Period following treatment with Placebo in the Double-blind Treatment Period.
- Cariprazine 3.0 mg/Day (Double-blind Safety Follow-up): Safety Follow-up Period following treatment with Cariprazine 3.0 mg/day in the Double-blind Treatment Period.
- Cariprazine 4.5 mg/Day (Double-blind Safety Follow-up): Safety Follow-up Period following treatment with Cariprazine 4.5 mg/day in the Double-blind Treatment Period.
Arm/Group | Cariprazine 4.5 mg/Day (Open-label Treatment Period) | Cariprazine 4.5 mg/Day (Open-label Safety Follow-up) | Placebo (Double-blind Treatment Period) | Cariprazine 3.0 mg/Day (Double-blind Treatment Period) | Cariprazine 4.5 mg/Day (Double-blind Treatment Period) | Placebo (Double-blind Safety Follow-up) | Cariprazine 3.0 mg/Day (Double-blind Safety Follow-up) | Cariprazine 4.5 mg/Day (Double-blind Safety Follow-up)
All-Cause Mortality (participants affected / at risk) | 1/587 | 0/273 | 0/54 | 0/49 | 0/56 | 0/54 | 0/49 | 0/56
Serious Adverse Events (participants affected / at risk) | 20/587 | 7/273 | 5/53 | 0/49 | 1/54 | 0/53 | 0/49 | 2/54
Other Adverse Events (participants affected / at risk) | 83/587 | 0/273 | 5/53 | 9/49 | 3/54 | 0/53 | 1/49 | 0/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cariprazine 4.5 mg/Day (Open-label Treatment Period) (N=587) | Cariprazine 4.5 mg/Day (Open-label Safety Follow-up) (N=273) | Placebo (Double-blind Treatment Period) (N=53) | Cariprazine 3.0 mg/Day (Double-blind Treatment Period) (N=49) | Cariprazine 4.5 mg/Day (Double-blind Treatment Period) (N=54) | Placebo (Double-blind Safety Follow-up) (N=53) | Cariprazine 3.0 mg/Day (Double-blind Safety Follow-up) (N=49) | Cariprazine 4.5 mg/Day (Double-blind Safety Follow-up) (N=54)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Schizophrenia (Psychiatric disorders) | 4 | 2 | 4 | 0 | 0 | 0 | 0 | 1
Delusion (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paranoia (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination, tactile (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Homicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Homicide (Social circumstances) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Miscarriage of partner (Social circumstances) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Social stay hospitalisation (Social circumstances) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract subcapsular (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0/188 | 1/95 | 0/14 | 0/17 | 0/22 | 0/14 | 0/17 | 0/22 — The number of participants at risk is based on the female population.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cariprazine 4.5 mg/Day (Open-label Treatment Period) (N=587) | Cariprazine 4.5 mg/Day (Open-label Safety Follow-up) (N=273) | Placebo (Double-blind Treatment Period) (N=53) | Cariprazine 3.0 mg/Day (Double-blind Treatment Period) (N=49) | Cariprazine 4.5 mg/Day (Double-blind Treatment Period) (N=54) | Placebo (Double-blind Safety Follow-up) (N=53) | Cariprazine 3.0 mg/Day (Double-blind Safety Follow-up) (N=49) | Cariprazine 4.5 mg/Day (Double-blind Safety Follow-up) (N=54)
Headache (Nervous system disorders) | 38 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 50 | 0 | 0 | 4 | 1 | 0 | 1 | 0
Cataract nuclear (Eye disorders) | 0 | 0 | 2 | 3 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 3 | 2 | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0/188 | 0/95 | 0/14 | 0/17 | 0/22 | 0/14 | 1/17 | 0/22 — Number of participants at risk is based on the female population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT03593213/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT03593213/SAP_001.pdf